CLINICAL TRIAL: NCT01108549
Title: Treatment of Chronic Fatigue Syndrome and Fibromyalgia With D-ribose- a Multicenter Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kona Research Center (Other)
Collaborators: Bioenergy Life Science, Inc. (Industry); Integrative Therapeutics, Inc. (Industry)
Responsible Party: Jacob Teitelbaum MD, Kona Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RiboseCFS03
Record Dates: First submitted 2010-04-16; First posted 2010-04-22 (Estimated); Last update posted 2010-04-22 (Estimated); Status verified 2010-04

CONDITIONS: Fibromyalgia; Chronic Fatigue Syndrome
Keywords: Fibromyalgia; Chronic Fatigue Syndrome; D-ribose; fatigue
MeSH Terms: conditions — Fibromyalgia; Fatigue Syndrome, Chronic; Fatigue | interventions — Ribose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Ribose — Ribose 5 grams PO TID was taken daily
  Other Names: D-ribose, corvalen

SUMMARY:
To determine whether adding Ribose 5 grams 3 x day would improve quality of life, energy, sleep and cognitive function and decrease pain in patients with CFS and/or fibromyalgia (CFS/FMS).

DETAILED DESCRIPTION:
Chronic Fatigue Syndrome and Fibromyalgia (CFS/FMS) are debilitating syndromes affecting ~ 2-4% of the population. Although they are heterogeneous conditions associated with many triggers, including infections, autoimmune illnesses, hormonal dysfunctions and other processes, they appear to have the common pathology of being associated with impaired energy metabolism.

As D-ribose has been shown to increase cellular energy synthesis in heart and skeletal muscle, and was shown to significantly improve clinical outcomes in CFS/FMS in an earlier pilot study, we conducted a larger, community based, multicenter trial to see if these findings could be generalized to a broader patient population. We hypothesized that giving D-ribose would improve function in CFS/FMS patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with Fibromyalgia (FMS) (by American College of Rheumatology [ACR] criteria) and/or Chronic Fatigue Syndrome (CFS- by Centers for Disease Control [CDC] criteria) by a health practitioner.

Exclusion Criteria:

* pregnant or nursing women, or
* any participants with known severe medication or nutrient sensitivities, or
* previous ribose use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2009-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
total score of hedonic scale of 5 symptoms | Change in total score of 5 symptoms after 3 weeks of treatment
  The assessed symptoms were energy, sleep, cognitive function, pain(inverse score) and overall sense of well being. Patients were asked to rate each of the 5 symptoms on a 1 to 7 scale

SECONDARY OUTCOMES:
Total of change in hedonic scale | at 1 week of treatment
  The assessed symptoms were energy, sleep, cognitive function, pain(inverse score) and overall sense of well being. Patients were asked to rate each of the 5 symptoms on a 1 to 7 scale
total change in hedonic scale | after 2 weeks of treatment
  The assessed symptoms were energy, sleep, cognitive function, pain(inverse score) and overall sense of well being. Patients were asked to rate each of the 5 symptoms on a 1 to 7 scale
Side effects | 3 weeks
  subjects and health practitioners were asked to report any side effects

CONTACTS AND LOCATIONS:
Overall Officials: Jacob E Teitelbaum, MD, Principal Investigator — Kona Research Center
Locations (1):
- Enzymatic Therapy, Green Bay, Wisconsin, United States